CLINICAL TRIAL: NCT02652819
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Efficacy and Safety of FG-4592 for Treatment of Anemia in Subjects With Chronic Kidney Disease Not on Dialysis
Brief Title: FG-4592 for Treatment of Anemia in Subjects With Chronic Kidney Disease Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-4592-808
Record Dates: First submitted 2015-12-31; First posted 2016-01-12 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Anemia
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FG-4592 (Experimental): Intervention is investigational treatment FG-4592
  Interventions: Drug: FG-4592
- Placebo (Placebo Comparator): Double blinded placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FG-4592
  Arms: FG-4592
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, multicenter, double-blind, placebo-controlled study of the treatment of anemia in subjects with CKD not on dialysis, with treatment up to 52 weeks.

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind, placebo-controlled study of the treatment of anemia in subjects with CKD not on dialysis.

Eligible subjects are randomized to FG-4592 or placebo at a ratio of 2:1. The primary endpoint is change in Hb from baseline to the average level during Weeks 7 to 9 inclusive.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75 years
2. Subject has voluntarily signed and dated an informed consent form (ICF), approved by an Ethics Committee (EC), after the nature of the study has been explained and the subject has had the opportunity to ask questions.
3. Diagnosis of chronic kidney disease, with Kidney Disease Outcomes Quality Initiative (KDOQI) Stage 3, 4, or 5, not receiving dialysis; with an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 estimated using the abbreviated 4-variable Modification of Diet in Renal Disease (MDRD) equation.
4. No use of an erythropoiesis-stimulating agent (ESA) for at least 5 weeks before randomization.
5. Mean of the two most recent Hb values during the Screening Period obtained at least 6 days apart must be ≥7.0 g/dL and <10 g/dL.
6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 x upper limit of normal (ULN), and normal total bilirubin at screening visit (based on central laboratory results).
7. Body weight: 40 to 100 kg inclusive.
8. Subjects agreeing not to start taking any new Traditional Chinese Medicine (TCM) for anemia and not to change dose, schedule, or brand of any prescreening TCM for anemia from beginning of Screening Period through end of Follow-up Period without approval of the FibroGen China Medical Monitor.

Exclusion Criteria:

1. Any clinically significant infection or evidence of an active underlying infection.
2. Positive for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus antibody (anti-HCV Ab).
3. Chronic liver disease.
4. New York Heart Association Class III or IV congestive heart failure.
5. Myocardial infarction, acute coronary syndrome, stroke, seizure, or a thromboembolic event (eg, deep venous thrombosis or pulmonary embolism) within 52 weeks prior to Day 1.
6. Uncontrolled hypertension in the opinion of the investigator (eg, that requires change in anti-hypertensive medication within 2 weeks prior to randomization).
7. Diagnosis or suspicion (eg, complex kidney cyst of Bosniak Category II or higher) of renal cell carcinoma as shown on screening renal ultrasound.
8. History of malignancy except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, or in situ cancer at any site.
9. Chronic inflammatory disease other than glomerulonephritis that could impact erythropoiesis (eg, systemic lupus erythematosis [SLE], rheumatoid arthritis, celiac disease).
10. Clinically significant gastrointestinal bleeding.
11. Known history of myelodysplastic syndrome, multiple myeloma, hereditary hematologic disease such as thalassemia, sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than CKD, hemosiderosis, hemochromatosis, known coagulation disorder, or hypercoagulable condition.
12. Any prior functioning organ transplant or a scheduled organ transplantation, or anephric.
13. Anticipated elective surgery that could lead to significant blood loss during the study period.
14. Anticipated use of dapsone or acetaminophen (paracetamol) >2.0 g/day, or >500 mg per dose repeated every 6 hours for more than 3 days.
15. Serum albumin <2.5 g/dL.
16. Androgen, deferoxamine, deferiprone, or deferasirox therapy within 12 weeks prior to Day 1.
17. Life expectancy of <12 months.
18. Blood transfusion within 12 weeks prior to Day 1 or anticipated need for transfusion.
19. IV iron supplement during the Screening Period and /or unwilling to withhold IV iron.
20. Immune suppressive or systematic steroid treatment within 12 weeks prior to Day 1.
21. History of alcohol or drug abuse within the past 2 years and inability to avoid consumption of more than >3 alcoholic beverages per day.
22. Prior treatment with FG-4592 or any hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI).
23. Use of an investigational medication or treatment, participation in an investigational interventional study, or carryover effect of an investigational treatment expected during the study.
24. Women who are pregnant or breastfeeding.
25. Women of childbearing potential and men with sexual partners of child bearing potential who are not using adequate contraception.
26. Any medical condition that, in the opinion of the investigator, may pose a safety risk to a subject in this study, may confound efficacy or safety assessment, or may interfere with study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01-24 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Change in Hb from baseline to the average level | Weeks 7 to 9 inclusive.
  Change in Hb from baseline to the average level

SECONDARY OUTCOMES:
The proportion of subjects who achieve a confirmed Hb response | up to and including Week 9
  The proportion of subjects who achieve a confirmed Hb response
Proportion of subjects with mean Hb ≥10.0 g/dL | Weeks 7 to 9
  Proportion of subjects with mean Hb ≥10.0 g/dL
Mean change from baseline in low-density lipoprotein (LDL) cholesterol averaged | Weeks 7 to 9
  Mean change from baseline in low-density lipoprotein (LDL) cholesterol averaged
Effect on iron metabolism | Week 9
  Measurement of serum iron
Survey (SF-36) Physical Functioning (PF) subscore measured in Week 9 in the Full Analysis Set (FAS) subjects with baseline PF subscore below 35 | Week 9
  Survey (SF-36) Physical Functioning (PF) subscore measured in Week 9 in the Full Analysis Set (FAS) subjects with baseline PF subscore below 35
Mean change from baseline in SF-36 vitality subscore measured in Week 9 in FAS subjects with baseline vitality subscore below 50. | Week 9
  Mean change from baseline in SF-36 vitality subscore measured in Week 9 in FAS subjects with baseline vitality subscore below 50.
Mean change from baseline in mean arterial blood pressure | Weeks 7 to 9
  Mean change from baseline in mean arterial blood pressure
Proportion of subjects who received rescue therapy (composite of blood transfusion, ESA use, and IV iron) | Up to Week 9
  Proportion of subjects who received rescue therapy (composite of blood transfusion, ESA use, and IV iron)
Percent of subjects with treatment-emergent adverse events (TEAEs). | Week 1 up to Week 53
  Percent of subjects with treatment-emergent adverse events (TEAEs) or serious adverse events (SAEs)
Number of subjects with treatment-emergent adverse events (TEAEs). | Week 1 up to Week 53
  Number of subjects with treatment-emergent adverse events (TEAEs) or serious adverse events (SAEs)
Changes from baseline in vital signs | Week 1 up to Week 53
  Measurement of vital signs
Changes from baseline in ECG findings | Week 1 up to Week 53
  ECG recordings
Changes from baseline in clinical laboratory values | Week 1 up to Week 53
  Clinical laboratory values
Proportion of subjects on rescue therapy | Week 1 up to Week 53
  Proportion of subjects on rescue therapy
Time to rescue therapy from date of first dose | Week 1 up to Week 53
  Time to rescue therapy from date of first dose

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - 301 Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Pekingg University, People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated hospital of Third Military Medical University (Southwest Hospital), Chongqing, Chongqing Municipality
  - Lan Zhou University Second Hospital, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated hospital of Guangxi Medical University, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of Baotou Medical School of Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medication, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medication, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan Universtiy, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Chen N, Hao C, Peng X, Lin H, Yin A, Hao L, Tao Y, Liang X, Liu Z, Xing C, Chen J, Luo L, Zuo L, Liao Y, Liu BC, Leong R, Wang C, Liu C, Neff T, Szczech L, Yu KP. Roxadustat for Anemia in Patients with Kidney Disease Not Receiving Dialysis. N Engl J Med. 2019 Sep 12;381(11):1001-1010. doi: 10.1056/NEJMoa1813599. Epub 2019 Jul 24. PMID 31340089